CLINICAL TRIAL: NCT06637774
Title: The Aspirometer: A Noninvasive Tool for Detecting Aspiration
Brief Title: The Aspirometer: A Noninvasive Tool for Detecting Aspiration Aim 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Toronto (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, James Coyle, Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: STUDY22040175 (Aim 3); R01HD074819 (NIH)
Record Dates: First submitted 2024-07-30; First posted 2024-10-15 (Actual); Results first posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Deglutition Disorders
Keywords: dysphagia; artificial intelligence; machine learning
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Prospective study of patients referred for videofluoroscopic swallow study, consenting to parallel data collection of signals. No control group.
Masking Description: Judges, examiners were blinded to participant diagnosis. Measurement/analysis judges were blinded to participant diagnosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Videofluoroscopic Swallow Study + Aspirometer (Experimental): Consecutively referred patients for modified barium swallow due to suspicion of dysphagia with aspiration, undergo the modified barium swallow test with Aspirometer sensors taped to the anterior neck. Signals are time-linked to images.
  Interventions: Device: Aspirometer; Device: Videofluoroscopic X-ray

INTERVENTIONS:
Device: Aspirometer — a triaxial accelerometer and a contact microphone affixed with tape to patient neck, a data accrual infrastructure, algorithms that decode swallow physiology noninvasively
  Other Names: high resolution cervical auscultation
Device: Videofluoroscopic X-ray — MBS is a fluoroscopic diagnostic test to evaluate swallowing physiology. Its images are judged by humans trained to do so.
  Other Names: Modified barium swallow study (MBS)

SUMMARY:
This investigation evaluates the effectiveness of a device called the Aspirometer, which uses high resolution cervical auscultation (HRCA), in detecting when food or liquids enter the airway (aspiration) of the person swallowing, whether the person swallowing shows signs of aspiration (coughing) or not.

DETAILED DESCRIPTION:
This aim of the project seeks to discriminate normal from abnormal airway protection and kinematic functions noninvasively via machine-learning analysis of Aspirometer/HRCA (high resolution cervical auscultation) signals, with similar accuracy as human judgment of VF. Hypothesis: Advanced data analytics can detect pathological airway protection in HRCA signal signatures with 90% accuracy when compared to a human expert's airway protection ratings from VF images. Analytical algorithms that can learn from data (e.g., Bayes' learning) will be used to infer about the continuum of abnormal airway protection during swallowing.

ELIGIBILITY:
Inclusion Criteria:

- referred by an attending physician as an inpatient, for a modified barium swallow examination due to suspected dysphagia and aspiration

Exclusion Criteria:

* tracheostomy
* pregnant
* unable to follow verbal commands
* anatomic disruption of head neck
* radiation therapy to head or neck

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Coyle, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center Oakland campus, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
algorithms, not individual participant data, will be made available to other researchers through an FTP (file transfer protocol) site

REFERENCES:
- [Background] Khalifa Y, Mahoney AS, Lucatorto E, Coyle JL, Sejdic E. Non-Invasive Sensor-Based Estimation of Anterior-Posterior Upper Esophageal Sphincter Opening Maximal Distension. IEEE J Transl Eng Health Med. 2023 Feb 20;11:182-190. doi: 10.1109/JTEHM.2023.3246919. eCollection 2023. PMID 36873304
- [Background] Mahoney AS, Khalifa Y, Lucatorto E, Sejdic E, Coyle JL. Cervical Vertebral Height Approximates Hyoid Displacement in Videofluoroscopic Images of Healthy Adults. Dysphagia. 2022 Dec;37(6):1689-1696. doi: 10.1007/s00455-022-10414-8. Epub 2022 Mar 1. PMID 35230537
- [Background] Schwartz R, Khalifa Y, Lucatorto E, Perera S, Coyle J, Sejdic E. A Preliminary Investigation of Similarities of High Resolution Cervical Auscultation Signals Between Thin Liquid Barium and Water Swallows. IEEE J Transl Eng Health Med. 2021 Dec 10;10:4900109. doi: 10.1109/JTEHM.2021.3134926. eCollection 2022. PMID 34963825
- [Background] Shu K, Coyle JL, Perera S, Khalifa Y, Sabry A, Sejdic E. Anterior-posterior distension of maximal upper esophageal sphincter opening is correlated with high-resolution cervical auscultation signal features. Physiol Meas. 2021 Apr 6;42(3). doi: 10.1088/1361-6579/abe7cb. PMID 33601360
- [Background] Donohue C, Khalifa Y, Perera S, Sejdic E, Coyle JL. A Preliminary Investigation of Whether HRCA Signals Can Differentiate Between Swallows from Healthy People and Swallows from People with Neurodegenerative Diseases. Dysphagia. 2021 Aug;36(4):635-643. doi: 10.1007/s00455-020-10177-0. Epub 2020 Sep 5. PMID 32889627
- [Background] Sejdic E, Malandraki GA, Coyle JL. Computational deglutition: Signal and image processing methods to understand swallowing and associated disorders. IEEE Signal Process Mag. 2019 Jan;36(1):138-146. doi: 10.1109/MSP.2018.2875863. Epub 2018 Dec 25. No abstract available. PMID 31631954
- [Background] Khalifa Y, Donohue C, Coyle JL, Sejdic E. Autonomous Swallow Segment Extraction Using Deep Learning in Neck-Sensor Vibratory Signals From Patients With Dysphagia. IEEE J Biomed Health Inform. 2023 Feb;27(2):956-967. doi: 10.1109/JBHI.2022.3224323. Epub 2023 Feb 3. PMID 36417738
- [Background] Donohue C, Khalifa Y, Mao S, Perera S, Sejdic E, Coyle JL. Characterizing Swallows From People With Neurodegenerative Diseases Using High-Resolution Cervical Auscultation Signals and Temporal and Spatial Swallow Kinematic Measurements. J Speech Lang Hear Res. 2021 Sep 14;64(9):3416-3431. doi: 10.1044/2021_JSLHR-21-00134. Epub 2021 Aug 24. PMID 34428093
- [Background] Donohue C, Khalifa Y, Mao S, Perera S, Sejdic E, Coyle JL. Establishing Reference Values for Temporal Kinematic Swallow Events Across the Lifespan in Healthy Community Dwelling Adults Using High-Resolution Cervical Auscultation. Dysphagia. 2022 Jun;37(3):664-675. doi: 10.1007/s00455-021-10317-0. Epub 2021 May 20. PMID 34018024
- [Background] Sabry A, Mahoney AS, Mao S, Khalifa Y, Sejdic E, Coyle JL. Automatic Estimation of Laryngeal Vestibule Closure Duration Using High- Resolution Cervical Auscultation Signals. Perspect ASHA Spec Interest Groups. 2020 Dec;5(6):1647-1656. doi: 10.1044/2020_persp-20-00073. Epub 2020 Dec 14. PMID 35937555
- [Background] Mao S, Sabry A, Khalifa Y, Coyle JL, Sejdic E. Estimation of laryngeal closure duration during swallowing without invasive X-rays. Future Gener Comput Syst. 2021 Feb;115:610-618. doi: 10.1016/j.future.2020.09.040. Epub 2020 Sep 30. PMID 33100445
- [Background] Coyle JL, Sejdic E. High-Resolution Cervical Auscultation and Data Science: New Tools to Address an Old Problem. Am J Speech Lang Pathol. 2020 Jul 10;29(2S):992-1000. doi: 10.1044/2020_AJSLP-19-00155. Epub 2020 Jul 10. PMID 32650655
- [Background] Khalifa Y, Coyle JL, Sejdic E. Non-invasive identification of swallows via deep learning in high resolution cervical auscultation recordings. Sci Rep. 2020 May 26;10(1):8704. doi: 10.1038/s41598-020-65492-1. PMID 32457331
- [Background] Donohue C, Mao S, Sejdic E, Coyle JL. Tracking Hyoid Bone Displacement During Swallowing Without Videofluoroscopy Using Machine Learning of Vibratory Signals. Dysphagia. 2021 Apr;36(2):259-269. doi: 10.1007/s00455-020-10124-z. Epub 2020 May 17. PMID 32419103
- [Background] Zhang Z, Perera S, Donohue C, Kurosu A, Mahoney AS, Coyle JL, Sejdic E. The Prediction of Risk of Penetration-Aspiration Via Hyoid Bone Displacement Features. Dysphagia. 2020 Feb;35(1):66-72. doi: 10.1007/s00455-019-10000-5. Epub 2019 Mar 27. PMID 30919104

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Videofluoroscopic Swallow Study + Aspirometer
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: adult inpatients referred for VFSS test due to suspected dysphagia
Arm/Group | Videofluoroscopic Swallow Study + Aspirometer
Number analyzed (Participants) | 50
Age, Continuous [Mean (Full Range); unit: years] | 66.77 [27.16 to 95.52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 46
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Numbers of Participants for Which the Aspirometer/HRCA Predicted the Passed Versus Failed Swallow Test Result
Description: Patients will undergo the Yale Swallow Protocol Screening Test and videofluoroscopic swallow study (VFS) while being concurrently monitored by the Aspirometer. Blinded trained human judges will score the screening test per its protocol indicating pass or fail based on the test's manual. Participants then immediately undergo a videofluoroscopic swallowing study during the same visit. Judgments of their penetration-aspiration scale (PAS) scores on the will serve as the gold standard for whether abnormal airway protection occurs during a swallow.
  The Yale swallow protocol involves a patient suspected of dysphagia with aspiration, drinking an aliquot of water (90mL) from a cup. Patient PASSES the screen if they drink the aliquot continuously without pausing, and if they do not cough or clear their throat after the swallow (one minute observation). Patients who PASS are assumed to NOT aspirate, patients who FAIL are assumed to aspirate.
Time Frame: day 1
Population: Only 23/50 patients produced single discrete swallows during VFS.
Measure: Count of Participants; unit: Participants
Arm/Group | Videofluoroscopic Swallow Study + Aspirometer
Number analyzed (Participants) | 23
Participants
  passed tests: number analyzed (Participants) | 5
  passed tests | 4
  failed tests: number analyzed (Participants) | 18
  failed tests | 12

2. Primary Outcome: Percentage of PAS Scores That Were Accurately Predicted by the Aspirometer/HRCA, in Comparison to Modified Barium Swallow Test.
Description: The Penetration Aspiration Scale is an 8-point ordinal scale validated in 1996. Scale range 1(best)-8(worst).
  Normal:
  1. no contrast entered the airway
  2. shallow laryngeal vestibule penetration of contrast above the vocal folds, NO airway residue observed
     Moderate:
  3. shallow laryngeal vestibule penetration above the vocal folds, airway residue IS observed
  4. deep laryngeal penetration to the inferior larynx, NO airway residue is observed
  5. deep laryngeal penetration to the inferior larynx, airway residue IS observed
  6. transient aspiration-contrast enters trachea and is ejected from trachea
     Severe:
  7. aspiration with observable tracheal residue, spontaneous airway clearance response ineffective
  8. silent aspiration-aspiration-no observed effort or reflexive reaction to clear airway
Time Frame: day 1
Measure: Count of Units; unit: PAS scores
Units Other Than Participants: PAS scores
Arm/Group | Videofluoroscopic Swallow Study + Aspirometer
Number analyzed (Participants) | 50
Number analyzed (PAS scores) | 85
PAS scores | 62

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Videofluoroscopic Swallow Study + Aspirometer
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/74/NCT06637774/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/74/NCT06637774/ICF_001.pdf